CLINICAL TRIAL: NCT05336513
Title: The Effect of an Anti-inflammatory Diet on Disease Activity and Quality of Life in Patients With Rheumatoid Arthritis - Parallel Controlled Randomized Clinical Trial
Brief Title: The Effect of an Anti-inflammatory Diet in Patients With Rheumatoid Arthritis
Acronym: DAIAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Nova de Lisboa (Other)
Collaborators: Hospital Particular do Algarve - HPA Saúde (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DAIAR
Record Dates: First submitted 2022-03-25; First posted 2022-04-20 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Rheumatoid Arthritis
Keywords: Anti-inflammatory diet; Disease activity; Quality of life; Rheumatoid arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diet Control (Other): Diet Control (DC): nutritional education and adherence monitoring. DC will be based on the Portuguese "Nova Roda dos Alimentos" following the principles of the Mediterranean diet.
  Interventions: Other: Diet Control
- Diet Anti-inflammatory (Experimental): Diet Anti-inflammatory (DAI): nutritional education and adherence monitoring. The DAI dietary intervention will be based on combining individual food items described as potential anti-inflammatory mitigators.
  Interventions: Other: Diet anti-inflammatory

INTERVENTIONS:
Other: Diet Control — Diet following mediterranean principles, for 15 weeks
  Arms: Diet Control
Other: Diet anti-inflammatory — Diet combining food items with anti-inflammatory potential, following the principles described in Rondanelli, Clinical Nutrition, 2021 Mar;40(3):661-689. doi: 10.1016/j.clnu.2020.08.020.
  Arms: Diet Anti-inflammatory

SUMMARY:
Rheumatoid arthritis (RA) is an autoimmune disease that affects 0.5-1% of the population and in which his remission is not always achieved, affecting physical and mental well-being and quality of life (QL). As a complement to pharmacotherapy, dietary intervention should be evaluated as a treatment option.

The main objective of this parallel controlled randomized clinical trial is to check the effect of an anti-inflammatory dietary intervention, compared to a diet based on the principles of the Mediterranean diet (control), on disease activity (AD) and improving QL.

Patients will be instructed to follow an anti-inflammatory diet (DAI) or a control diet (DC) for 6 months. The AD and QL will be evaluated at the end of the intervention.

As there are no dietary guidelines for RA, this study aims to provide scientific evidence about the impact of diet therapy on reducing AD and improving QL.

DETAILED DESCRIPTION:
The main objective of this trial is to check the effect of an DAI, compared to a DC, on reducing AD and improving QL.

As secondary objectives, it is intended to investigate the relationship of DAI with inflammatory markers and with the modulation of the composition / diversity of the intestinal microbiota, in comparison with a DC.

This study combines all dietary components with an anti-inflammatory effect, thus allowing the possibility of evaluating the full potential of dietary treatment in the disease, including intestinal microbiota modulation.

These results are intended to further contribute to clinical decision making and better evidence-based treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years;
* Presence of active disease, (DAS28≥ 2.6), under adequate control and medication.
* Able to sign informed consent

Exclusion Criteria:

* Any type of psychological deficiency, dementia or eating disorder;
* Presence of food allergies and / or intolerances;
* Be vegetarian or use Phytotherapy or other supplements (namely, pre and probiotics);
* Use of antibiotics im the last 6 months;
* Have had previous nutritional monitoring or change in eating habits in the last 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
Changes in disease activity | 15 weeks
  Difference between the intervention and control group in the changes in Disease Activity (using DAS28 score: greater than 2,6 implies active disease), from baseline to the end of follow-up
Changes in Quality of Life | 15 weeks
  Difference between the intervention and control group in changes in Quality of Life (Health Assessment Questionnaire (HAQ): scores of 0 to 1 are generally considered to represent mild to moderate difficulty, 1 to 2 moderate to severe disability, and 2 to 3 severe to very severe disability), from baseline to the end of follow-up

SECONDARY OUTCOMES:
Changes in C-Reactive Protein (CRP) | 15 weeks
  Difference between the intervention and control group in changes in C-Reactive Protein (CRP) measured in mg/L, from baseline to the end of follow-up
Changes in Erythrocyte Sedimentation Rate (ESR) | 15 weeks
  Difference between the intervention and control group in changes in Erythrocyte Sedimentation Rate (ESR) measured in mm/h, from baseline to the end of follow-up
Changes in Rheumatoid Factor (RF) | 15 weeks
  Difference between the intervention and control group changes in Rheumatoid Factor (RF) measured in IU/mL, from baseline to the end of follow-up
Changes in Gut microbiota | 15 weeks
  Difference between the intervention and control group in the change of gut microbiota from baseline to the end of follow-up.
  Bacterial DNA will be extracted from fecal samples. 16SRNA gene will be sequenced by next-generation sequencing (NGS). All the identified bacterial phyla, genus and species will be expressed in percentage.
Changes in weight | 15 weeks
  Difference between the intervention and control group changes in weight, measured in Kg, from baseline to the end of follow-up
Changes in Body Mass Index (BMI) | 15 weeks
  Difference between the intervention and control group changes in BMI, calculated using weight and height, presented in kg/m2: underweight < 18,5; normoweight 18,6-24,9; overweight 25-29,9; obese >30, from baseline to the end of follow-up
Changes in waist circumference perimeter | 15 weeks
  Difference between the intervention and control group changes in waist circumference perimeter, measured in cm, from baseline to the end of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Ana Faria, PhD, Principal Investigator — Universidade Nova de Lisboa
Locations (1):
- Hospital Particular do Algarve - HPA Saúde, Portimão, Portugal

IPD SHARING:
Plan to Share IPD: Undecided